CLINICAL TRIAL: NCT06022237
Title: Efficacy and Safety of Oral Ibandronate in Patients of Liver Cirrhosis With Hepatic Osteodystrophy: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Efficacy and Safety of Oral Ibandronate in Patients of Liver Cirrhosis With Hepatic Osteodystrophy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-61
Record Dates: First submitted 2023-08-22; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hepatic Osteodystrophy; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Ibandronic Acid; Calcium; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibandronate (Experimental): Ibandronate 150 mg once monthly in a supervised manner in front of student investigator and will be observed for 2 hours following ingestion. Patients will also receive Calcium 500mg BD and Vitamin D3 1000 mg OD
  Interventions: Drug: Ibandronate; Drug: Calcium; Drug: Vitamin D3
- Placebo (Active Comparator): Group B will receive placebo once monthly along with Calcium 500mg BD and Vitamin D3 1000 mg OD
  Interventions: Drug: Calcium; Drug: Vitamin D3

INTERVENTIONS:
Drug: Ibandronate — Ibandronate 150 mg once monthly.
  Arms: Ibandronate
Drug: Calcium — Calcium 500 mg twice daily
Drug: Vitamin D3 — Vitamin D3 - 1000 IU daily

SUMMARY:
Hepatic osteodystrophy(HOD) is a common but frequently overlooked complication of liver cirrhosis with a prevalence rate ranging from 13-70%. Bisphosphonates acting by inhibiting bone resorption are frequently used. Intravenous infusions of bisphosphonates may cause prolonged arthralgia and myalgia whereas oral bisphosphonates may cause digestive mucosal damage causing dysphagia, esophagitis and ulcer. Such side effects have discouraged the prescription of oral bisphosphonates for patients of cirrhosis mainly due to risk of upper GI hemorrhage arising from esophageal variceal rupture.

All studies done in past with bisphosphonates are either open labelled RCT/ non- randomized control trial or have enrolled patients of primary biliary cirrhosis only.

So, there is a need to have double blind RCT assessing efficacy and safety of oral bisphosphonates in non-cholestatic liver cirrhosis.

In this study, we hypothesize that oral ibandronate significantly improves BMD in patients of liver cirrhosis & is safe in patients with low risk esophageal varices. With this study, we aim to assess the efficacy and safety of oral ibandronate in patients of liver cirrhosis with hepatic osteodystrophy

DETAILED DESCRIPTION:
Hypothesis : Oral ibandronate 150 mg once monthly significantly improves BMD in patients of liver cirrhosis with hepatic osteodystrophy by decreasing bone resorption & is safe in patients with low risk esophageal varices.

Methodology:

Study population: All the consecutive patients with liver cirrhosis attending department of Hepatology will be evaluated for inclusion criteria. The diagnosis of cirrhosis will be confirmed either by liver biopsy or associated clinical, radiological and endoscopic findings compatible with cirrhosis and PH.

All enrolled patients will undergo detailed evaluation by thorough history ,clinical examination and relevant laboratory investigations.

All cirrhotic patients will be subjected to upper GI endoscopy. Patients with low risk esophageal varices(grade I and II without red-color signs) and low risk GOV-1/GOV2 will be subjected to DEXA scan to measure BMD at femur neck and lumbar spine. Patient with grade II and III varices with RCS will be enrolled only after EVL after 6-8 weeks until varices achieve a low risk status described as eradicated/grade I & II varices without RCS

Patients with HOD (osteoporosis according to WHO criteria :BMD T score< -2.5) or with osteopenia(BMD T score between -1 and -2.5) will be enrolled in our study

Informed consent will be taken from all patients.

Study design: Prospective double blind randomized control trial

Study period: 1 year Sample size: 80

Our primary objective is to compare changes in BMD (delta T) at lumbar spine in DEXA scan after 1 year of oral ibandronate therapy. As shown by Guanabens N et al. Hepatology 2013 Dec;58(6):2070-8) that assuming baseline T score in both groups(Ibandronate & placebo) were comparable & after 1 year the mean T score increased by 0.393 i.e delta T of 0.393 in bisphosphonate group & delta T of 0.1 in placebo group, we need to enroll 68 cases i.e 34 in each group with alpha error of 5% & power 95%. Further assuming defaulter rate of 20%, it is decided to enroll 80 cases i.e 40 in each group randomly allocated into 2 groups by block randomization method taking block size of 8.

Intervention: All enrolled patients will be randomly allocated into 2 groups by block randomization method taking block size of 8.

Group A will receive Ibandronate 150 mg once monthly in a supervised manner in front of student investigator and will be observed for 2 hours following ingestion. Group A will also receive Calcium and Vitamin D3. Group B will receive placebo once monthly along with Calcium and Vitamin D3

Monitoring and assessment:

Group A will receive Ibandronate 150 mg once monthly in fasting state with a glass of water in sitting posture and the patient will be instructed to not to lie down or eat for at least 30 minutes. Contact number of student investigator will be given to the patient to report symptoms in the next 48 hours. .Patient will be asked to maintain diary to report and monitor symptoms and inform student investigator

CBC ,KFT, LFT, PT/INR, HBsAg, HCV, ANA, ASMA, Anti-LKM, Ceruloplasmin and iron studies will be carried out in all enrolled patients at the time of enrollment. USG abdomen will be performed in all cases and triple phase CT of abdomen when there will be suspicion of HCC. Serum calcium, phosphate,25(OH)D, Fasting thyroid profile and PTH level will also be estimated.

Following four biochemical markers of bone turnover will be tested at entry and end of study:

* Serum osteocalcin,
* PICP( procollagen type 1 C propeptide)
* NTX (aminoterminal cross-linking telopeptide of type I collagen)
* CTX (carboxyterminal cross-linking telopeptide of type I collagen)

Lateral radiograph of thoracic and lumbar spine will be obtained at entry and after 1 year in all patients to disclose fracture rates in both groups. Vertebral fracture will be defined as reduction of >20 % in the anterior, middle or posterior height of vertebral body. Fracture attributable to major trauma will not be recorded. Development of new peripheral fracture due to trivial trauma will also be monitored All patients will be followed every month and oral ibandronate will be given in a supervised manner under observation of student investigator for 2 hours.

Biochemical bone turnover marker and DEXA scan will be repeated after 1 year of follow up. LFT and Liver fraility index will be assessed every 3 month. Upper GI endoscopy will be repeated at the end of study and as when required.

Adverse effects: Patients may be made aware of the possible side effects of the study drug. During each follow up visit, patient will be thoroughly evaluated for any side effects of ibandronate: UGI bleed, dyspeptic symptoms, and musculoskeletal symptoms (myalgia/arthralgia).Only complaints within 48 hours of taking medicine that limit daily activities will be documented.

Stopping rule: Patient experiencing UGI bleed, dyspeptic symptoms, and musculoskeletal symptoms (myalgia/arthralgia) within 48 hours of oral ibandronate, intractable dyspeptic symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis patients between 18 to 70 yrs with low risk esophageal varices and HOD (osteoporosis/osteopenia will be enrolled).
2. Patient and attendants willing to give informed consent

Exclusion Criteria:

1. Age <18 years and > 70 years
2. Patients with prior history of fracture
3. History of upper GI bleed in last 2 months
4. Patients with post EVL ulcers
5. High risk esophageal varices or gastric varices without endoscopic treatment.
6. Active peptic ulcer
7. Severe vascular ectasia
8. Esophageal stricture
9. Achalasia
10. Creatinine clearance below 30ml/min
11. Malignancy(except HCC)
12. Hyperparathyroidism
13. Patients using NSAIDs, corticosteroids ,anticoagulants or ongoing alcohol beverages
14. Bisphosphonate hypersensitivity/Oral bisphosphonate within 12 months
15. Grade 2/3 ascites
16. Hepatic encephalopathy(Grade 3 &4)
17. Critically ill patients
18. Post LT patients
19. HRT within 6 mths
20. Pregnant and lactating women
21. Patient with bleeding disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMD at lumbar spine | 1 year

SECONDARY OUTCOMES:
Change in BMD at femur neck | 1 year
Incidence of UGI bleed in both arms | 1 year
Change in bone turnover marker after 1 year of ibandronate | 1 year
Association between T-score of DEXA scan at lumbar spine and femur neck with (Child-Turcotte-Pugh (CTP) score. | 1 year
Association between T-score of DEXA scan at lumbar spine and femur neck with Model for End Stage Liver Disease score. | 1 year
Fracture rate after 1 year of ibandronate therapy | 1 year
Change in liver fraility index after 1 year of ibandronate therapy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No